CLINICAL TRIAL: NCT03434301
Title: Comparison of Mesh Fixation Techniques in Elective Laparoscopic Repair of Incisional Hernia - ReliaTack™ v ProTack™ (TACKoMesh Study)
Brief Title: Comparison of Mesh Fixation Techniques in Elective Laparoscopic Repair of Incisional Hernia - ReliaTack™ v ProTack™
Acronym: TACKoMesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R04484
Record Dates: First submitted 2018-01-29; First posted 2018-02-15 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Incisional Hernia; Hernia; Abdominal Hernia
Keywords: Surgery; Laparotomy; Tack; Non-absorbable Tack; Absorbable Tack; Pain
MeSH Terms: conditions — Incisional Hernia; Hernia; Hernia, Abdominal; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesh with absorbable tack fixation (Active Comparator): Mesh with absorbable tack (ReliaTack™) fixation
  Interventions: Device: ReliaTack™
- Mesh with non-absorbable fixation (Active Comparator): Mesh with non-absorbable (Protack™) fixation
  Interventions: Device: Protack™

INTERVENTIONS:
Device: ReliaTack™ — Absorbable tack (ReliaTack™) to fixate Symbotex™ composite mesh in the elective repair of incisional hernia.
  Arms: Mesh with absorbable tack fixation
Device: Protack™ — Non-absorbable tack (Protack™) to fixate Symbotex™ composite mesh in the elective repair of incisional hernia.
  Arms: Mesh with non-absorbable fixation

SUMMARY:
This study is designed to examine the effects on post operative pain after the use of a fixation device to secure a mesh in the abdomen to repair a hernia of the abdominal wall. The fixation devices to be used differ with one being made from titanium and is permanent and the other being made from an absorbable material. Both fixation devices are commonly used but two questions remain unanswered, does one cause more chronic pain and also what if any will be the effect on recurrence rates of the hernia. No trial has been undertaken to date which will not only examine the fixation device but in the setting where the hernia is closed first. The closure of the hernial defect by the keyhole technique is a relatively new and growing concept in the hernia world.

DETAILED DESCRIPTION:
TACKoMESH study (Comparison of using absorbable tacks (ReliaTack™) against a non-absorbable tack (Protack™) to fixate Symbotex™ composite mesh in the elective repair of incisional hernia) is a prospective, single-centre, double blinded randomised trial which aims to establish whether the use of absorbable (ABS) compared to non-absorbable (Non-ABS) tacks in adult patients undergoing elective incisional hernia repair produces a lower rate of pain both immediately and long-term. Secondary outcomes to be explored include seroma formation, hernia recurrence, length of postoperative hospital stay, wound infection, reoperation rate, operation time, health related quality of life and time to return to normal daily activity.

Patients entering TACKoMesh will be randomised immediately prior to their operation with a 1:1 ratio of ABS versus Non-ABS tack arm allocation. The same composite mesh will be used for all operations. Follow-up is according to a predetermined schedule, using specifically designed Case Report Forms to collect the blinded data.

ELIGIBILITY:
Inclusion Criteria:

• All adults undergoing elective incisional hernia repair for midline abdominal incisional hernia, with a defect of 3-10cm in diameter.

Exclusion Criteria:

* Patients less than 18 years of age, or unable to give informed consent.
* Patients over 80 years of age.
* Females of reproductive age.
* Prisoners.
* Clinically small incisional hernia <3cm maximum diameter.
* Emergency procedures (for irreducible, strangulated or obstructed hernia).
* Procedure involving dirty (purulent inflammation (e.g. abscess); preoperative perforation of respiratory, gastrointestinal, biliary or genitourinary tract; penetrating trauma >4 hours old) or contaminated (Non-purulent inflammation; gross spillage from gastrointestinal tract; entry into biliary or genitourinary tract in the presence of infected bile or urine; major break in technique; penetrating trauma <4 hours old; chronic open wounds to be grafted or covered) surgery.
* Patients with a Body Mass Index (BMI) >40 kg/m².
* Patients participating in any other study, whose concurrent participation in the TACK study might place them at undue risk or might confound the study data in the opinion of the chief investigators.
* Failure to close the anterior rectus sheath intraoperatively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Pain score | 30 days
  Pain Score at rest and activity at day 30 recorded using visual analogue pain score (VAS) (0-10cm).

SECONDARY OUTCOMES:
Visual analogue pain score (VAS). | Day 1, days 5-7, 3 months, 1 year.
  Visual analogue pain score (VAS) pain score at days 1, 5-7 3 months and 1 year post-operative. A preoperative VAS score will also be recorded.
Seroma formation. | Days 1, 6, 30, 3 months and 1 year post-operation.
  Seroma formation (no fixed time point) (a seroma will be defined as any clinically apparent fluid collection at the site of mesh placement).
Postoperative hospital stay. | Time from end of Surgery to patient discharge (up to end of study; 104 weeks).
  The length of postoperative hospital stay.
Time to return to normal daily activity. | From day of surgery to end of study (104 weeks).
  The time to return to normal daily activity.
Wound infection. | Days 1, 6, 30, 3 months and 1 year post-operation.
  Any wound infection.
Operating time. | Length of Operation.
  The time taken for the Operation - from start to finish.
Mesh fixation time. | Time during Operation.
  Mesh fixation time after adhesions have been taken down and fascia closed.
Hernia recurrence. | Days 1, 6, 30, 3 months and 1 year post-operation.
  Hernia recurrence at one year and at all time points.
Health-related quality of life. | 30 days and 1 year post-operation.
  Health-related quality of life - assessed using the Carolinas Comfort Score™ (which is specifically designed for hernia repair) (26) and Short Form 36™, at pre-operatively, 30 days and 1 year, (appendix K and SF-36).
Adverse Events. | Days 1, 6, 30, 3 months and 1 year post-operation.
  To capture any Adverse Events during the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Aali J Sheen, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheen AJ, Pilkington JJ, Baltatzis M, Tyurkylmaz A, Stathakis P, Jamdar S, Siriwardena AK. Comparison of Mesh Fixation Techniques in Elective Laparoscopic Repair of Incisional Hernia-ReliaTack v ProTack (TACKoMesh) - A double-blind randomised controlled trial. BMC Surg. 2018 Jul 11;18(1):46. doi: 10.1186/s12893-018-0378-3. PMID 29996841